CLINICAL TRIAL: NCT00232466
Title: VERTOS II. Percutaneous Vertebroplasty Versus Conservative Therapy in Patients With Osteoporotic Vertebral Fractures
Brief Title: VERTOS-II. Percutaneous Vertebroplasty Versus Conservative Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Office Imaging Division (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor-Investigator, Clinical Research Office Imaging Division, Clinical research coordinator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 945-06-351; 945-06-351
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2008-06

CONDITIONS: Osteoporosis; Back Pain
Keywords: Vertebroplasty; Vertebral fracture; Actonel; Osteoporotic; vertebral; fractures
MeSH Terms: conditions — Osteoporosis; Back Pain; Spinal Fractures; Fractures, Bone | interventions — Vertebroplasty

ARMS (2):
- 2 (No Intervention): conservative therapy (no intervention)
- 1 (Active Comparator): Vertebroplasty
  Interventions: Procedure: Vertebroplasty

INTERVENTIONS:
Procedure: Vertebroplasty — Procedure:
  The treatment consists of a transpedicular injection of polymethylmethacrylate bone cement into the collapsed vertebral body (maximal 2 vertebrae in 1 treatment session) using fluoroscopic guidance. The procedure is performed under the use of local anesthetics and the patient can be discharged the same day or after 1 night of hospital stay.
  Arms: 1

SUMMARY:
Percutaneous vertebroplasty is a new procedure for treating painful osteoporotic compression fractures of the spine. Five-thousand out of 12.000 patients (16.000 vertebral fractures/year in the Netherlands) present with sudden, severe back pain in the region of the fracture.Until recently, bed rest, analgesia and physical support were the only treatment options. After decades of performing PV, no large RCT with mid-term follow-up has been published.

Design:

This will be a multicenter (6 centers), prospective, randomised, intervention study. Eligible patients will be randomised for percutaneous vertebroplasty or conservative therapy.

Study population:

Age: 50 and older, vertebral fracture, level: thoracic vertebral body 5 (Th 5) or lower, osteopenia (T-score < -1 SD), back pain for no more than 6 weeks and edema in the vertebrae on MR imaging

Statistical analyses All analyses will be performed on an 'intention to treat' principle. The planned number of subjects will be 200 in total, 100 in each intervention arm.

Economic evaluation:

Cost-effectiveness will be assessed. The costs of the procedure and the medical treatment, and of visits to medical specialists, GP's and physical therapists will be compared.

Time schedule:

The total study will take 36 months

Recruitment of patients (200) has been completed. In May 2009 the 1 year follow-up will be finished.

DETAILED DESCRIPTION:
Design:

This will be a multicenter (6 centers), prospective, randomized, intervention study. Eligible patients will be randomized for percutaneous vertebroplasty or analgesics.

Study population:Two hundred patients will be included.

Patient selection:

Patients will be referred from the GP to the radiology department for acute back pain. The GP will order an X-ray of the thoracic and lumbar spine to establish an osteoporotic vertebral fracture(s). Subsequently, the hospital radiologist will pick out the cases with vertebral fracture(s). Subsequently, the general physician/ geriatrician will confirm the diagnosis of 'osteoporotic' vertebral fracture, and exclude other causes of vertebral fracture (e.g. tumour, major trauma). Finally, the patient and their GP will be asked to participate in our study.

Eligible patients will be randomized for percutaneous vertebroplasty (and pain medication if necessary) or only analgesics.

Procedure:

The treatment consists of a transpedicular injection of polymethylmethacrylate bone cement into the collapsed vertebral body (maximal 2 vertebrae in 1 treatment session) using fluoroscopic guidance. The procedure is performed under the use of local anesthetics and the patient can be discharged the same day or after 1 night of hospital stay.

Conventional treatment (analgesics):

The internist optimizes the use of analgesics in ascending order: (1) Paracetamol, (2) Tramadol, (3) Tramadol and Paracetamol, (4) Morphine.

All patients receive osteoporosis medication.

Outcome parameters:

The primary outcome for the clinical study as well as the economic evaluation will be adequate relief of pain. Pain intensity will be measured by means of a visual analogue scale (VAS). Relief of up to 3,0 to 4,4 scale points (scale 0-10) is associated with a clinically relevant pain reduction (Beurskens et al 1995). The main goal of the economic evaluation is to assess the balance between costs and effects of percutaneous vertebroplasty and pain medication as compared to usual care (analgesics, physiotherapy, visits to general practitioner) after 4 weeks and after 1 year.

The clinical research objectives are to compare the effects (1 day,1 week, 1 month, 3 months, 6 months,12 months and 24 months) of vertebroplasty with conventional therapy on a) back pain, b) activities of daily living (ADL), c) mood, d) general health and e) quality of life in patients with painful osteoporotic vertebral fractures. Other objectives are to study the 1 and 2-year incidence of recurrent fractures, especially adjacent to treated levels of

Measurements:

a), b), c), d) and e) are measured by using the visual analogue scale (VAS) for pain intensity, the Roland Disability Questionnaire (RDQ) for functional status, while, the EQ6D and the Qualeffo-41 focus on quality of life, mood and general health. Data will be collected about units of resource utilization with an explicit clause asking whether it can be related to the vertebral fracture.

(New) osteoporotic vertebral fractures are assessed at baseline by conventional radiography and magnetic resonance (MR) imaging. The incidence of recurrent fractures will be determined by conventional X-rays at 1,3,12 and 24 months.

Economic evaluation:

The goal of the economic evaluation is to assess the balance between costs and effects of vertebroplasty as compared to usual care.

We will initially perform a cost-effectiveness analysis with a one month time horizon. Given immediate pain relief in a majority after vertebroplasty, already a cost-effectiveness ratio can be calculated.

Estimates of other relevant outcomes such as costs and quality of life will also be entered in the model to allow a full economic evaluation. We will estimate incremental costs per additional year freed of pain of immediate vertebroplasty as compared to vertebroplasty after one month and (synthetic scenario of) care as usual. As the latter does involve extrapolation using estimates not actually observed in the trial we can not use bootstrap simulation to assess uncertainty. Accordingly, multivariate probabilistic sensitivity analysis (Monte carlo simulations) will be used to evaluate uncertainty in the cost-effectiveness ratios. As we will take into account a time horizon up till one year costs nor effects will be discounted. Finally, a cost-utility analysis is foreseen based on utility scores obtained over the first month of observation after randomization.

The direct medical costs will be estimated from a societal perspective. This implies that resource use such as GP visits, analgesics, physiotherapy and consultation of orthopedic surgeons or general physicians will be recorded in the CRF and in patient diaries. In parallel, actual costs of the resources, i.e., unit costs, will be estimated. The majority will be based on the estimates gathered in the Dutch guidelines for economic evaluation published by CVZ. Subsequently, multiplication of units costs with resource use will yield cost estimates on an individual patient level. With regard to costs due to losses in productivity we pose that the majority of patients does not have a paid job. Time spent by spouses, family and friends taking over certain household activities or other unpaid activities will be accounted for using shadow prices.

The primary outcome for the economic evaluation will be adequate relief of pain. Pain will be measured by means of a visual analogue scale (VAS). Relief of up to 3,0 to 4,4 scale points is considered adequate. Time until this outcome is attained will explicitly be accounted for in the economic evaluation.

In addition to pain, health related quality of life will be measured. Subsequent summation over the period of follow up will yield overall QALYs up to a year for each arm of the trial.

In the cost effectiveness analysis we will take care of the differences in the Belgium and Dutch healthcare system.

Statistical analyzes All analyzes will be performed on an intention to treat principle. In addition, analyzes will on the different outcomes will be compared between the two groups with the Student's t-test for continuous normally distributed variables, with the Mann-Whitney test for variables that are not normally distributed and with the chi² test for categorical variables. In addition, subgroups (e.g. long/shot duration of complaints) will be examined in which vertebroplasty has a more (or less) pronounced effect by introducing interaction terms in linear regression models with change in pain and quality of life as outcome variables.

The one-year cumulative incidence of new fractures adjacent to the treated/old fracture levels will be compared between patients who were treated with vertebroplasty and those who were not with Cox-proportional hazards analyzes, adjusting for confounders.

Power calculations:

The planned number of subjects will be 200 in total, 100 in each intervention arm. This number is based on conventional assumptions of alfa=0.05 and ß=0.20, withdrawal from intervention of 20%. Based on pilot data and literature we expect a difference of 25% in significant pain relief. If we assume that 20% withdraws from intervention we need approximately 100 patients in each group.

Time schedule:

The total study will take 36 months.

Recruitment of patients (200) has been completed. In May 2009 the 1 year follow-up will be finished.

ELIGIBILITY:
Inclusion criteria:

* age: 50 and older
* vertebral fracture: 15-85% height loss
* level: thoracic vertebral body 5 (Th 5) or lower
* osteopenia (T-score < -1 SD)
* back pain for at least no longer than 6 weeks
* edema in the vertebrae on MR imaging

Exclusion criteria:

* complete loss of vertebral body height
* fracture through or destruction of the posterior vertebral wall
* pressure of bone fragments on the spinal cord
* osteomyelitis or spondylodiscitis
* vertebral column neoplasms
* uncorrectable coagulation disorder
* medical conditions that would make the patient ineligible for emergency decompressive surgery should it be necessary to treat a complication of the procedure

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-02; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To compare the cost-effectivity in the two groups | 1 month, 1 year
VAS score in time | 1 month, 1 year

SECONDARY OUTCOMES:
To compare pain relief and the quality of life of the patients in the two groups. | 1 day, 1 week, 1 month, 3 months, 6 months, 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Willem Mali, MD.PhD, Principal Investigator — UMC Utrecht
Locations (6):
- AZ St. Lucas Ziekenhuis, Ghent, Belgium
- Netherlands (5):
  - Diakonessenhuis, Utrecht/Zeist/Doorn, Utrecht
  - Albert Schweizer Ziekenhuis, Dordrecht
  - Catharina-Ziekenhuis, Eindhoven
  - St. Elisabeth Ziekenhuis, Tilburg
  - UMCU, Utrecht

REFERENCES:
- [Derived] Klazen CA, Lohle PN, de Vries J, Jansen FH, Tielbeek AV, Blonk MC, Venmans A, van Rooij WJ, Schoemaker MC, Juttmann JR, Lo TH, Verhaar HJ, van der Graaf Y, van Everdingen KJ, Muller AF, Elgersma OE, Halkema DR, Fransen H, Janssens X, Buskens E, Mali WP. Vertebroplasty versus conservative treatment in acute osteoporotic vertebral compression fractures (Vertos II): an open-label randomised trial. Lancet. 2010 Sep 25;376(9746):1085-92. doi: 10.1016/S0140-6736(10)60954-3. Epub 2010 Aug 9. PMID 20701962
- [Derived] Klazen CA, Venmans A, de Vries J, van Rooij WJ, Jansen FH, Blonk MC, Lohle PN, Juttmann JR, Buskens E, van Everdingen KJ, Muller A, Fransen H, Elgersma OE, Mali WP, Verhaar HJ. Percutaneous vertebroplasty is not a risk factor for new osteoporotic compression fractures: results from VERTOS II. AJNR Am J Neuroradiol. 2010 Sep;31(8):1447-50. doi: 10.3174/ajnr.A2148. Epub 2010 Jul 22. PMID 20651016
- [Derived] Venmans A, Klazen CA, Lohle PN, van Rooij WJ, Verhaar HJ, de Vries J, Mali WP. Percutaneous vertebroplasty and pulmonary cement embolism: results from VERTOS II. AJNR Am J Neuroradiol. 2010 Sep;31(8):1451-3. doi: 10.3174/ajnr.A2127. Epub 2010 May 20. PMID 20488908
- [Derived] Klazen CA, Verhaar HJ, Lampmann LE, Juttmann JR, Blonk MC, Jansen FH, Tielbeek AV, Schoemaker MC, Buskens E, van der Graaf Y, Janssens X, Fransen H, van Everdingen KJ, Muller AF, Mali WP, Lohle PN. VERTOS II: percutaneous vertebroplasty versus conservative therapy in patients with painful osteoporotic vertebral compression fractures; rationale, objectives and design of a multicenter randomized controlled trial. Trials. 2007 Oct 31;8:33. doi: 10.1186/1745-6215-8-33. PMID 17973983
- See also: information about vertebroplasty — http://www.vertebroplastiek.nl